CLINICAL TRIAL: NCT04727294
Title: Monoclonal Gammopathy of Undetermined Significance (MGUS), Smoldering Myeloma (SMM), and Multiple Myeloma Patient Experience With COVID-19 Survey
Brief Title: MGUS, SMM, and MM Patient Experience With Coronavirus 19 (COVID-19) Survey
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: HealthTree Foundation (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: MM/COVID-19 part II
Record Dates: First submitted 2021-01-26; First posted 2021-01-27 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-08

CONDITIONS: Multiple Myeloma; Smoldering Multiple Myeloma; Monoclonal Gammopathy of Undetermined Significance; Coronavirus
Keywords: Questionnaire
MeSH Terms: conditions — Multiple Myeloma; Smoldering Multiple Myeloma; Monoclonal Gammopathy of Undetermined Significance; Coronavirus Infections | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MGUS, SMM, MM Patients or their Caregivers: Eligible participants will be asked to create a free patient profile on the HealthTree Cure Hub (www.healthtree.org) or use their existing patient profile.
  The creation of a HealthTree Cure Hub patient profile will serve as a screen for eligibility.
  Patients will complete a one-time questionnaire found on the HealthTree Cure Hub. Telephone assistance can be provided as needed. The questionnaire will take 20-30 minutes to complete.
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Series of questions covering COVID-19 diagnosis and treatment, changes in myeloma treatment and care, clinical trial familiarity, health and fitness, and quality of life.

SUMMARY:
The purpose of this study is to examine how patients with multiple myeloma (MM) have been impacted by the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) pandemic.

The study will use a questionnaire to further understand how patients are being affected and gather information in order to track the long-term effects of the coronavirus.

The scope of the questionnaire will include, COVID-19 diagnosis and treatment, changes in myeloma treatment and care, clinical trial familiarity, health and fitness, and quality of life.

This questionnaire is a follow-on to the "MM and COVID-19" questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (greater than 18 years) diagnosed with MGUS, smoldering myeloma, and multiple myeloma.
* Access to a computer or electronic device with internet access, or phone
* Willing to create a patient profile on the HealthTree Cure Hub For Multiple Myeloma
* Willing to give electronically-signed consent
* Ability to read questions in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with MGUS, smoldering myeloma, or multiple myeloma.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2021-01-22 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
COVID-19 Diagnosis and Treatment | Up to one year
  Describe how patients diagnosed with COVID-19 were treated for the virus.
Changes to Myeloma Treatment and Care | Up to one year
  Describe which treatments were changed and how care was affected as a result of COVID-19
Health and Fitness | Up to one year
  Describe how COVID-19 impacted patient's health and fitness
Quality of Life (QOL) Distress Screening tool | Up to one year
  Describe how patients rate their level of concern on psychosocial, practical, and physical needs during the COVID-19 pandemic using the Cancer Support Community's CancerSupportSource distress screening tool.

SECONDARY OUTCOMES:
Clinical Trial Familiarity | Upon enrollment
  Describe how familiar patients are with multiple myeloma clinical trials.

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Sweeney, PhD, Study Chair — HealthTree Foundation
Locations (1):
- HealthTree.org (Online), Lehi, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
The HealthTree foundation values responsible and ethical sharing of data from clinical trials. De-identified patient responses to the questionnaire will be aggregated and shared back with the patient. Additionally, portions of the de-identified results will be shared with the research community through publications (abstracts, reports, manuscripts).
Supporting Information: Study Protocol, ICF, CSR
Access Criteria: Visit the HealthTree Foundation's online patient portal: HealthTree Cure Hub For Multiple Myeloma
URL: http://healthtree.org